CLINICAL TRIAL: NCT00447759
Title: Phase 4 Study A Large Streamline Safety Study Designed to Compare the Cardiovascular Safety od Celecoxib Versus Traditional Non-selective NSAID's
Brief Title: The Standard Care Versus Celecoxib Outcome Trial
Acronym: SCOTLSSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: University of Glasgow (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCOT Trial
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
Keywords: Celecoxib; Celebrex; Ibuprofen; Diclofenac; NSAID; Osteoarthritis; Rheumatoid Arthritis; Arthritis; Safety study; Cardiovascular safety; Clinical trial; PROBE design; University of Dundee; Medicines Monitoring Unit; MEMO; Professor Tom MacDonald
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis | interventions — Celecoxib; Diclofenac; Ibuprofen; Naproxen; Meloxicam

STUDY DESIGN:
Intervention Model Description: Prospective Randomised Open Blinded-Endpoint Study (PROBE)
Masking Description: NSAID
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Celecoxib (Experimental): Celecoxib. Celebrex 200-400mg daily in divided doses
  Interventions: Drug: Celecoxib
- Diclofenac (Active Comparator): continue usual nsNSAID
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Celecoxib — 200-400mg daily in divided doses
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Diclofenac — prescribed medication taken orally
  Other Names: Ibuprofen; Naproxen; meloxicam; other presribed sNSAIDs
  Arms: Diclofenac

SUMMARY:
The Standard Care versus Celecoxib Outcome Trial (SCOT) is a large streamline safety study designed to compare the cardiovascular safety of celecoxib versus traditional non-selective Non Steroidal Anti-Inflammatory Drug (NSAID) therapy.Traditional NSAID's are associated with significant morbidity and mortality from gastrointestinal toxicity. Cyclooxygenase 2 (Cox-2)selective agents are associated with reduced upper gastrointestinal toxicity.Traditional NSAID's and Cox-2 inhibitors may also be associated with cardiovascular and renal disorders. Data from both randomised and observational studies suggest that celecoxib has similar or reduced cardiovascular toxicity when compared to traditional NSAID's. However, the overall safety balance of a strategy of celecoxib therapy versus a strategy of NSAID therapy is unknown. The European Medicines Evaluation Agency (EMEA) has requested that studies of the cardiovascular safety of celecoxib be carried out within the indicated population of Europe. This study addresses these issues by comparing the cardiovascular safety of celecoxib therapy with traditional NSAID therapy in the setting of the EU healthcare system.

As of May 2013, 7300 patients had been randomised, and had accrued an average 4.2 years of follow up by the end of May 2014.

DETAILED DESCRIPTION:
Aims

The present proposal seeks to compare the cardiovascular and gastrointestinal safety and effectiveness of a strategy of initial randomisation to treatment with the selective COX-2 inhibitor celecoxib or to 'usual-care' with their current non-selective NSAID therapy (with or without cyto-protection with ulcer healing drug use in either celecoxib or 'usual-care' limbs).

Trial Design

This trial utilises the Prospective Randomised Open Blinded End point (PROBE) design . Patients with clinically diagnosed osteoarthritis (OA) or rheumatoid arthritis (RA) 60 years of age or more who are free from established cardiovascular disease and who require chronic NSAID therapy will be identified in the setting of primary care. Patients will be randomised to receive either celecoxib or to continue their previous standard NSAID therapy. They will then be followed up for an average of 4.2 years in the setting of the local National Healthcare system. The study will terminate when 277 adjudicated cardiovascular events have accrued. A summary is shown in the diagram below.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 60 years or over Male & Female
* Chronic NSAIDs use for 90 days or more in a 12 month period
* Subjects who have a licensed indication for chronic non-selective NSAID or Celecoxib.
* Eligible for treatment with either Celecoxib or alternative traditional non-selective NSAID.
* Subjects who are willing to consent to their paper and electronic medical records and prescribing data to be accessed.
* Subjects who are willing to be contacted and interviewed by trial investigators.

Exclusion Criteria:

* Established cardiovascular disease including ischaemic heart disease, Myocardial Infarction, angina or acute coronary syndrome, cerebrovascular disease or cerebrovascular accident or transient ischaemic attack, established peripheral vascular disease and moderate to severe heart failure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7297 (Actual)
Dates: Start 2007-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
compare cardiovascular safety of celecoxib and traditional NSAIDs prescribed for the treatment of arthritis. | 4 years

SECONDARY OUTCOMES:
demonstrate the superiority of celecoxib over traditional NSAIDs on ulcer-related upper gastrointestinal complications. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M MacDonald, MD MRCP FRCP, Principal Investigator — University of Dundee; Ian Ford, FRCP FRSE, Principal Investigator — University of Glasgow; Christopher J Hawkey, MRCP DM FRC, Principal Investigator — University of Nottingham
Locations (10):
- University of Southern Denmark, Odense, Denmark
- Julius Clinical Research, Zeist, Netherlands
- United Kingdom (8):
  - University of Aberdeen, Aberdeen
  - University of Birmingham, Birmingham
  - University of Dundee, Dundee
  - University of Edinburgh, Edinburgh
  - University of Glasgow, Glasgow
  - NHS Highlands, Inverness
  - University of Nottingham, Nottingham
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Data released on application to steering committee
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 28/08/2015
Access Criteria: Open Access Journals
URL: https://www.dundee.ac.uk/memo/

REFERENCES:
- [Background] MacDonald TM. A European's perspective of COX-2 drug safety. J Cardiovasc Pharmacol. 2006;47 Suppl 1:S92-7. doi: 10.1097/00005344-200605001-00017. PMID 16785838
- [Derived] MacDonald TM, Hawkey CJ, Ford I, McMurray JJV, Scheiman JM, Hallas J, Findlay E, Grobbee DE, Hobbs FDR, Ralston SH, Reid DM, Walters MR, Webster J, Ruschitzka F, Ritchie LD, Perez-Gutthann S, Connolly E, Greenlaw N, Wilson A, Wei L, Mackenzie IS. Randomized trial of switching from prescribed non-selective non-steroidal anti-inflammatory drugs to prescribed celecoxib: the Standard care vs. Celecoxib Outcome Trial (SCOT). Eur Heart J. 2017 Jun 14;38(23):1843-1850. doi: 10.1093/eurheartj/ehw387. PMID 27705888
- [Derived] Jennings CG, MacDonald TM, Wei L, Brown MJ, McConnachie L, Mackenzie IS. Does offering an incentive payment improve recruitment to clinical trials and increase the proportion of socially deprived and elderly participants? Trials. 2015 Mar 7;16:80. doi: 10.1186/s13063-015-0582-8. PMID 25888477
- [Derived] Macdonald TM, Mackenzie IS, Wei L, Hawkey CJ, Ford I; SCOT study group collaborators. Methodology of a large prospective, randomised, open, blinded endpoint streamlined safety study of celecoxib versus traditional non-steroidal anti-inflammatory drugs in patients with osteoarthritis or rheumatoid arthritis: protocol of the standard care versus celecoxib outcome trial (SCOT). BMJ Open. 2013 Jan 29;3(1):e002295. doi: 10.1136/bmjopen-2012-002295. PMID 23364320